CLINICAL TRIAL: NCT04417218
Title: Determinants of Alpha-aminoadipic Acid (2-AAA) and Relationship to Diabetes: Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jane Ferguson, Assistant Professor, Cardiovascular Medicine Division, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200427; R01DK117144 (NIH)
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — Lysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Lysine Diet (Experimental): Participants will complete two one-week dietary interventions, in a randomized order. For the normal lysine diet, participants will be asked to adhere to a specific diet for 1 week. Each study subject will receive 3 meals and 1-2 snacks per day during the study period.
  Interventions: Dietary Supplement: Controlled Diet
- High Lysine Diet (Experimental): Participants will complete two one-week dietary interventions, in a randomized order. For the high lysine diet, participants will be asked to consume the same foods as in the normal lysine diet, but with the addition of lysine supplements (5g/day).
  Interventions: Dietary Supplement: Lysine; Dietary Supplement: Controlled Diet

INTERVENTIONS:
Dietary Supplement: Lysine — Lysine is an essential amino acid which is acquired from dietary sources.
  Arms: High Lysine Diet
Dietary Supplement: Controlled Diet — Individuals will be instructed to consume specific foods, to adhere to a controlled lysine diet.

SUMMARY:
This study aims to assess the effect of controlled dietary lysine intake on plasma and urine α-aminoadipic acid (2-AAA).

DETAILED DESCRIPTION:
Diabetes is an important health concern worldwide. It is associated with significantly increased mortality as well as high incidence of co-morbidities. Unfortunately, treatment efficacy and successful disease management is highly variable among treated patients, and this is partly due to the fact that diabetes has multiple underlying causes most of which are still unknown. A newly identified biomarker, α-aminoadipic acid (2-AAA), has the potential to successfully predict the development of diabetes in humans, even before the development of other known risk markers. However, little is known about the function of 2-AAA; it is unclear whether 2-AAA itself causes the development of diabetes or if it is a biomarker for altered metabolic processes that then lead to diabetes.

The aim of the first phase of the study was to measure plasma 2-AAA levels from healthy individuals from the general population to identify subjects with high or low 2-AAA. Now in the second phase of the study, 80 subjects with high or low 2-AAA will be invited to participate in a dietary lysine modification study to access the effect of controlled lysine intake on plasma and urine 2AAA. Participants will be asked to complete two one-week dietary interventions. Subjects will be screened and consented via email, online, or phone. Each subject will be required to come to Vanderbilt University Medical Center for four study visits, at which the study team will obtain a blood sample, a urine sample, stool sample, vital signs, waist and hip circumference, and 1-3 surveys will be completed if the subject did not complete them prior to the visit. Each subject that completes the entire study visit will be compensated $250. DNA samples will be obtained to allow for identification of genetic predictors of 2-AAA levels. Some individuals may be asked to return for a future follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Prior participant in 2-AAA screening study.
* Identified as eligible due to high or low plasma 2-AAA, in the absence of hyperglycemia, as defined by study team.

Exclusion Criteria:

* Individuals who currently use tobacco products.
* Use of prescription or over-the-counter medications or dietary supplements which could modulate levels of 2-AAA and unwilling to discontinue use (from 24 hours prior to first study visit until completion of study). Hormonal birth control is acceptable.
* Follow a severely restricted diet or have food allergies, which would preclude adherence to study diet.
* Newly diagnosed disease (since screening visit), including cardiovascular, renal, or liver disease, or Diabetes mellitus.
* Individuals who are pregnant or lactating
* Inability to provide written or electronic informed consent
* Inability to fast for 8 hours

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: N=20 enrolled individuals withdrew or were lost to follow up prior to starting the intervention.
Groups:
- Normal Lysine Diet First Then High Lysine Diet: Participants completed two one-week dietary interventions, in a randomized order, separated by a 2-week washout.
  For the Normal Lysine diet, participants were asked to adhere to a specific diet for 1 week. Individuals were instructed to consume specific foods, to adhere to a controlled lysine diet. This comprised 3 meals and 1-2 snacks per day during the study period.
  For the Washout, individuals were asked to resume their habitual diet for 2 weeks.
  For the High Lysine diet, participants were asked to adhere to a specific diet for 1 week. Individuals were instructed to consume the same specific foods, as the Normal Lysine diet. This comprised 3 meals and 1-2 snacks per day during the study period. Participants were also instructed to take Lysine supplements with their meals (5g/day).
  Lysine: Lysine is an essential amino acid which is acquired from dietary sources.
  Controlled Diet: Individuals will be instructed to consume specific foods, to adhere to a controlled lysine diet.
- High Lysine Diet First Then Normal Lysine Diet: Participants completed two one-week dietary interventions, in a randomized order, separated by a 2-week washout.
  For the High Lysine diet, participants were asked to adhere to a specific diet for 1 week. Individuals were instructed to consume specific foods. This comprised 3 meals and 1-2 snacks per day during the study period. Participants were also instructed to take Lysine supplements with their meals (5g/day).
  For the Washout, individuals were asked to resume their habitual diet for 2 weeks.
  For the Normal Lysine diet, participants were asked to adhere to a specific diet for 1 week. Individuals were instructed to consume specific foods (the same as during the High Lysine diet), to adhere to a controlled lysine diet. This comprised 3 meals and 1-2 snacks per day during the study period.
  Lysine: Lysine is an essential amino acid which is acquired from dietary sources.
  Controlled Diet: Individuals will be instructed to consume specific foods, to adhere to a controlled lysine diet.
Period: First Intervention (1 Week))
Arm/Group | Normal Lysine Diet First Then High Lysine Diet | High Lysine Diet First Then Normal Lysine Diet
Started | 25 | 22
Completed | 24 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Normal Lysine Diet First Then High Lysine Diet | High Lysine Diet First Then Normal Lysine Diet
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Normal Lysine Diet First Then High Lysine Diet | High Lysine Diet First Then Normal Lysine Diet
Started | 24 | 22
Completed | 24 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dietary Intervention: Participants will complete two one-week dietary interventions, in a randomized order. For the normal lysine diet, participants will be asked to adhere to a specific diet for 1 week. Each study subject will receive 3 meals and 1-2 snacks per day during the study period.
  Controlled Diet: Individuals will be instructed to consume specific foods, to adhere to a controlled lysine diet.
  For the high lysine diet, participants will be asked to consume the same foods as in the normal lysine diet, but with the addition of lysine supplements (5g/day).
  Lysine: Lysine is an essential amino acid which is acquired from dietary sources.
Arm/Group | Dietary Intervention
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma 2-AAA Concentration From Baseline
Description: Alpha aminoadipic acid (2-AAA) concentration determined through mass spectrometry, quantified to standard. The change was calculated as post-diet minus pre-diet for each Intervention (Normal lysine and High lysine).
Time Frame: Change from pre-diet to post-diet (1 week)
Population: Individuals were included for analysis only if they had provided a blood sample for measurement of 2-AAA at both the pre- and post-diet timepoints. This excluded 3 individuals from the normal lysine diet intervention, and 4 individuals from the high lysine diet intervention.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Normal Lysine Diet | High Lysine Diet
Number analyzed (Participants) | 43 | 42
ng/ml | -9.35 (30.3) | 7.02 (23.7)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected over the 4 week study period.
Arm/Group | Normal Lysine Diet | High Lysine Diet
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 2/47 | 7/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normal Lysine Diet (N=47) | High Lysine Diet (N=46)
Bloating (Gastrointestinal disorders) | 1 (1) | 4 (4) — Reports of bloating, gas, or GI discomfort
Changes in mood (Psychiatric disorders) | 0 (0) | 1 (1) — reported improvement in mood
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Change in mood (Psychiatric disorders) | 0 (0) | 1 (1) — reported nervousness
Bruising (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Reported pain and bruising following blood draw.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT04417218/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04417218/ICF_000.pdf